CLINICAL TRIAL: NCT03070951
Title: A Phase 3, Multicentre, Randomized, Double-blind, Placebo-controlled Study Investigating the Efficacy and Safety of Daily Oral Administration of OBE2109 Alone and in Combination With Add-back Therapy for the Management of Heavy Menstrual Bleeding Associated With Uterine Fibroids in Premenopausal Women
Brief Title: Efficacy and Safety of OBE2109 in Subjects With Heavy Menstrual Bleeding Associated With Uterine Fibroids
Acronym: PRIMROSE 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ObsEva SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-OBE2109-009
Record Dates: First submitted 2017-02-17; First posted 2017-03-06 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Uterine Fibroids; Heavy Menstrual Bleeding
Keywords: Uterine Fibroid; Leiomyomata; Heavy Menstrual Bleeding; HMB; Heavy Uterine Bleeding; Menorrhagia; OBE2109 + Add-back
MeSH Terms: conditions — Leiomyoma; Menorrhagia | interventions — linzagolix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- OBE2109 dose 1 (100mg) + Placebo Add-back (Experimental)
  Interventions: Drug: OBE2109; Drug: Placebo to match OBE2109; Drug: Placebo to match Add-back
- OBE2109 dose 1 (100mg) + Add-back (Experimental)
  Interventions: Drug: OBE2109; Drug: Placebo to match OBE2109; Drug: Add-back
- OBE2109 dose 2 (200mg) + Placebo Add-back / OBE2109 dose 2 (200 mg) + Add-back (Experimental)
  Interventions: Drug: OBE2109; Drug: Placebo to match Add-back; Drug: Add-back
- OBE2109 dose 2 (200mg) + Add-back (Experimental)
  Interventions: Drug: OBE2109; Drug: Add-back
- Placebo + Placebo Add-back / OBE2109 dose 3 (200mg) + Add-back (Placebo Comparator)
  Interventions: Drug: OBE2109; Drug: Placebo to match OBE2109; Drug: Placebo to match Add-back; Drug: Add-back

INTERVENTIONS:
Drug: OBE2109 — OBE2109 100mg tablets for oral administration once daily
Drug: Placebo to match OBE2109 — Placebo to match OBE2109 100mg tablets for oral administration once daily
  Arms: OBE2109 dose 1 (100mg) + Add-back; OBE2109 dose 1 (100mg) + Placebo Add-back; Placebo + Placebo Add-back / OBE2109 dose 3 (200mg) + Add-back
Drug: Placebo to match Add-back — Placebo to match Add-back (E2 1 mg / NETA 0.5 mg) for oral administration once daily
  Arms: OBE2109 dose 1 (100mg) + Placebo Add-back; OBE2109 dose 2 (200mg) + Placebo Add-back / OBE2109 dose 2 (200 mg) + Add-back; Placebo + Placebo Add-back / OBE2109 dose 3 (200mg) + Add-back
Drug: Add-back — Add-back (E2 1 mg / NETA 0.5 mg) for oral administration once daily
  Arms: OBE2109 dose 1 (100mg) + Add-back; OBE2109 dose 2 (200mg) + Add-back; OBE2109 dose 2 (200mg) + Placebo Add-back / OBE2109 dose 2 (200 mg) + Add-back; Placebo + Placebo Add-back / OBE2109 dose 3 (200mg) + Add-back

SUMMARY:
The primary objective of this study is to demonstrate the superior efficacy versus placebo of OBE2109 alone and in combination with add-back therapy for the reduction of heavy menstrual bleeding associated with uterine fibroids in premenopausal women.

DETAILED DESCRIPTION:
The study is a prospective, randomized, parallel group, double-blind, placebo-controlled phase 3 study investigating the efficacy and safety of OBE2109 alone and in combination with add-back therapy for the treatment of uterine fibroids.

Subjects will be randomized to one of 5 treatment groups in a 1:1:1:1:1 ratio.

ELIGIBILITY:
Key Inclusion Criteria:

* Premenopausal woman at screening.
* Body Mass Index ≥ 18 kg/m2.
* Menstrual cycles ≥ 21 days and ≤ 40 days.
* Presence of uterine fibroids.
* Heavy menstrual blood loss for each of the 2 menstrual periods assessed at screening using the alkaline hematin method.

Key Exclusion Criteria:

* The subject is pregnant or breast-feeding or is planning a pregnancy within the duration of the treatment period of the study.
* History of uterus surgery that would interfere with the study.
* The subject's condition is so severe that she will require surgery within 6 months regardless of the treatment provided.
* Undiagnosed abnormal uterine bleeding.
* Significant risk of osteoporosis or history of, or known osteoporosis or other metabolic bone disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 511 (Actual)
Dates: Start 2017-05-23 (Actual); Primary Completion 2019-09-16 (Actual); Study Completion 2020-10-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Responders based on menstrual blood loss (MBL) volume reduction at Week 24 | From baseline to Week 24
  Assessed using the alkaline hematin method

SECONDARY OUTCOMES:
Time to reduced menstrual blood loss | Up to Week 52
  Assessed using the alkaline hematin method
Amenorrhea | Up to Week 52
  Assessed using the alkaline hematin method
Time to amenorrhea | Up to Week 52
Number of days of uterine bleeding for the last 28-day interval prior to Week 24 | last 28-day interval prior to Week 24
  Assessed using the alkaline hematin method
Number of days of uterine bleeding for each 28-day interval | Up to Week 52
  Assessed using the alkaline hematin method

OTHER OUTCOMES:
Bone Mineral Density (BMD) | From baseline up to Week 76
  Assessed by dual-energy X-ray absorptiometry (DXA) scan
Endometrial biopsy | From baseline up to Week 52
  Assessed by histology
Adverse events | Up to Week 76
  Frequency and severity of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: ObsEva SA, Study Director — Geneva
Locations (96):
- United States (23):
  - Site reference ID 905, Chino, California
  - Site reference ID 918, Huntington Park, California
  - Site reference ID 902, San Diego, California
  - Site reference ID 903, Denver, Colorado
  - Site reference ID 913, Bradenton, Florida
  - Site reference ID 912, Orlando, Florida
  - Site reference ID 915, Augusta, Georgia
  - Site reference ID 924, Nampa, Idaho
  - Site reference ID 926, Covington, Louisiana
  - Site reference ID 927, Metairie, Louisiana
  - Site reference ID 900, Metairie, Louisiana
  - Site reference ID 901, Canton, Michigan
  - Site reference ID 932, Detroit, Michigan
  - Site reference ID 916, Jefferson City, Missouri
  - Site reference ID 930, Albuquerque, New Mexico
  - Site reference ID 933, West Seneca, New York
  - Site reference ID 931, Hamlet, North Carolina
  - Site reference ID 914, Westerville, Ohio
  - Site reference ID 928, Erie, Pennsylvania
  - Site reference ID 919, West Columbia, South Carolina
  - Site reference ID 907, Houston, Texas
  - Site reference ID 911, Salt Lake City, Utah
  - Site reference ID 917, Madison, Wisconsin
- Bulgaria (11):
  - Site reference ID 265, Gabrovo
  - Site reference ID 255, Pleven
  - Site reference ID 258, Plovdiv
  - Site reference ID 266, Sliven
  - Site reference ID 264, Smolyan
  - Site reference ID 251, Sofia
  - Site reference ID 252, Sofia
  - Site reference ID 254, Sofia
  - Site reference ID 256, Sofia
  - Site reference ID 257, Sofia
  - Site reference ID 267, Sofia
- Czechia (9):
  - Site reference ID 285, České Budějovice
  - Site reference ID 283, Písek
  - Site reference ID 281, Prague
  - Site reference ID 286, Prague
  - Site reference ID 287, Prague
  - Site reference ID 288, Prague
  - Site reference ID 284, Příbram
  - Site reference ID 289, Tábor
  - Site reference ID 282, Vsetín
- Hungary (9):
  - Site reference ID 315, Baja
  - Site reference ID 303, Budapest
  - Site reference ID 307, Budapest
  - Site reference ID 301, Debrecen
  - Site reference ID 308, Debrecen
  - Site reference ID 313, Debrecen
  - Site reference ID 314, Kecskemét
  - Site reference ID 304, Kistarcsa
  - Site reference ID 306, Nyíregyháza
- Latvia (3):
  - Site reference ID 451, Riga
  - Site reference ID 452, Riga
  - Site reference ID 454, Riga
- Lithuania (4):
  - Site reference ID 463, Kaunas
  - Site reference ID 460, Vilnius
  - Site reference ID 461, Vilnius
  - Site reference ID 464, Vilnius
- Poland (17):
  - Site reference ID 502, Bialystok
  - Site reference ID 504, Katowice
  - Site reference ID 509, Katowice
  - Site reference ID 513, Katowice
  - Site reference ID 514, Katowice
  - Site reference ID 501, Knurów
  - Site reference ID 510, Lodz
  - Site reference ID 517, Lodz
  - Site reference ID 506, Lublin
  - Site reference ID 508, Lublin
  - Site reference ID 511, Lublin
  - Site reference ID 519, Piaseczno
  - Site reference ID 518, Poznan
  - Site reference ID 505, Przemyśl
  - Site reference ID 503, Szczecin
  - Site reference ID 512, Świdnik
  - Site reference ID 507, Warsaw
- Romania (5):
  - Site reference ID 606, Brasov
  - Site reference ID 601, Bucharest
  - Site reference ID 603, Bucharest
  - Site reference ID 604, Bucharest
  - Site reference ID 605, Târgu Mureş
- Ukraine (15):
  - Site reference ID 813, Chernivtsi
  - Site reference ID 801, Ivano-Frankivsk
  - Site reference ID 814, Kharkiv
  - Site reference ID 802, Kyiv
  - Site reference ID 803, Kyiv
  - Site reference ID 805, Kyiv
  - Site reference ID 806, Kyiv
  - Site reference ID 807, Kyiv
  - Site reference ID 804, Lviv
  - Site reference ID 811, Odesa
  - Site reference ID 808, Ternopil
  - Site reference ID 817, Vinnytsia
  - Site reference ID 812, Zaporizhzhya
  - Site reference ID 815, Zaporizhzhya
  - Site reference ID 816, Zaporizhzhya

REFERENCES:
- [Derived] Donnez J, Petraglia F, Taylor H, Becker CM, Becker S, Herrera FC, Bestel E, Hori S, Dolmans MM. Linzagolix with and without hormonal add-back therapy for symptomatic uterine fibroids: PRIMROSE 1 & 2 long-term extension and withdrawal study. Fertil Steril. 2025 Oct;124(4):737-748. doi: 10.1016/j.fertnstert.2025.06.016. Epub 2025 Jun 19. PMID 40543832
- [Derived] Becker S, Dolmans MM, Herrera FC, Petraglia F, Renner SP, Ionescu-Ittu R, St-Pierre J, Boolell M, Bestel E, Hori S, Donnez J. Pain Reduction in Linzagolix-Treated Patients With Uterine Fibroids: A Secondary Mediation Analysis of the PRIMROSE 1 and 2 Phase 3 Trials. BJOG. 2025 Aug;132(9):1297-1306. doi: 10.1111/1471-0528.18190. Epub 2025 May 6. PMID 40326221
- [Derived] Donnez J, Taylor HS, Stewart EA, Bradley L, Marsh E, Archer D, Al-Hendy A, Petraglia F, Watts N, Gotteland JP, Bestel E, Terrill P, Loumaye E, Humberstone A, Garner E. Linzagolix with and without hormonal add-back therapy for the treatment of symptomatic uterine fibroids: two randomised, placebo-controlled, phase 3 trials. Lancet. 2022 Sep 17;400(10356):896-907. doi: 10.1016/S0140-6736(22)01475-1. PMID 36116480